CLINICAL TRIAL: NCT02814422
Title: Triglyceride-rich Lipoprotein and the Development of Dementia
Brief Title: Triglyceride-rich Lipoprotein and Development of Dementia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201407002RIND
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Dementia
Keywords: Triglyceride-rich lipoprotein; dementia; Alzheimer's disease; mild cognition impairment; amyloid-beta
MeSH Terms: conditions — Dementia; Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Because of the rapid aging of the global population, dementia has become a serious problem, and Alzheimer's disease (AD) is the most common cause of dementia. AD is pathologically characterized by substantial neuronal loss and chronic inflammation that is associated with cerebrovascular and parenchymal accumulation of proteinaceous deposits enriched in amyloid-beta (Aβ). More recent evidence shows it is due to an increased blood-to-brain delivery of circulating Aβ, and significant peripheral Aβ metabolism occurs in association with post-prandial triglyceride-rich lipoproteins.

In the prodromal stage of AD, patients usually suffer mild cognition impairment (MCI). The annual conversion rate of MCI to AD is around 10%, and within 3 years, around 30%-50% of these develop dementia. Brain atrophy is an irreversible brain disease that causes problems with cognitive and memory functions in many diseases, such as MCI and AD, etc. In order to allow preventive intervention for AD, MCI must be diagnosed as early as possible, using biomarker assays or simple imaging modality. From 2009-2013, the investigators have registered 4,492 patients with atherosclerotic vascular diseases (AVD). In addition, the investigators have also registered 8,209 cases with no evidence of AVD, but with at least 1 cardiovascular risk factor. In this 5-year project, 300 male or female patients with stable symptomatic AVD over 20 years of age, and the other 600 patients with no evidence of AVD but with at least 1 CV risk factor, will be enrolled from our previous registry program. The baseline and yearly follow-up study will include clinical examination, neurocognitive function evaluation, and laboratory tests (TC, HDL-C, LDL-C, TG, hs-CRP, and Aβ-40, Aβ-42, tau protein, and other biological signatures: adiponectin, MMP-3, MMP-9, IL-6, Fibrinogen, Lp-PLA2, 8-Isoprostane, hFABP, sVCAM-1, sICAM-1, CA-125, MCP-1, TNF-α, cTnI, NT-proBNP, CNP, NGAL).

The purposes of this 5-year project are (1) to clarify the association of triglyceride-rich lipoprotein and the development of dementia; (2) to validate the diagnostic power and prognostic implication of ultra-low-concentration biomarkers (Aβ-40, Aβ-42 and tau) for dementia.

DETAILED DESCRIPTION:
Because of the rapid aging of the global population, dementia has become a serious problem, and Alzheimer's disease (AD) is the most common cause of dementia. Population studies have shown that dietary fats influence risk and progression of age-related diseases including AD, diabetes and cardiovascular disease. Consumption of saturated fat, trans-fatty acids and cholesterol are positively associated with increased risk. These findings support the hypothesis that dietary saturated-fats (SFA) and cholesterol, or dietary induced dyslipidemia are causally associated with AD risk. AD is pathologically characterized by substantial neuronal loss and chronic inflammation that is associated with cerebrovascular and parenchymal accumulation of proteinaceous deposits enriched in amyloid-beta (Aβ). More recent evidence shows it is due to an increased blood-to-brain delivery of circulating Aβ, and significant peripheral Aβ metabolism occurs in association with post-prandial triglyceride-rich lipoproteins.

In the prodromal stage of AD, patients usually suffer mild cognition impairment (MCI). The annual conversion rate of MCI to AD is around 10%, and within 3 years, around 30%-50% of these develop dementia. Brain atrophy is an irreversible brain disease that causes problems with cognitive and memory functions in many diseases, such as MCI and AD, etc. In order to allow preventive intervention for AD, MCI must be diagnosed as early as possible, using biomarker assays or simple imaging modality. From 2009-2013, the investigators have registered 4,492 patients with atherosclerotic vascular diseases (AVD). In addition, the investigators have also registered 8,209 cases with no evidence of AVD, but with at least 1 cardiovascular risk factor. In this 5-year project, 300 male or female patients with stable symptomatic AVD over 20 years of age, and the other 600 patients with no evidence of AVD but with at least 1 CV risk factor, will be enrolled from our previous registry program. The baseline and yearly follow-up study will include clinical examination, neurocognitive function evaluation, and laboratory tests (TC, HDL-C, LDL-C, TG, hs-CRP, and Aβ-40, Aβ-42, tau protein, and other biological signatures: adiponectin, MMP-3, MMP-9, IL-6, Fibrinogen, Lp-PLA2, 8-Isoprostane, hFABP, sVCAM-1, sICAM-1, CA-125, MCP-1, TNF-α, cTnI, NT-proBNP, CNP, NGAL).

ELIGIBILITY:
Inclusion Criteria:

* age older than 20 years old
* willing to sign ICF
* report oneself disease
* have Taiwanese ID
* atherosclerotic vascular diseases, but with at least 1 CV risk factor [DM, dyslipidemia or under lipid lowering therapy, hypertension, smoking, old (M>45, F>55 years), family history of premature CAD, obesity

Exclusion Criteria:

* not willing to sign ICF

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In this project, three hundred male or female patients with stable symptomatic atherosclerotic disease over 20 years of age will be enrolled from our previous registry program. Peripheral atherosclerosis with symptoms of ischemia and confirmed by ankle-brachial index, Doppler ultrasound, or angiography will also be included (group A). The other 1000 patients will be enrolled with no evidence of atherosclerotic vascular diseases, but with at least 1 CV risk factor [DM, dyslipidemia (TC >200 mg/dL; LDL-C > 130 mg/dL ; TG > 200 mg/dL; male HDL-C < 40 mg/dL ; female HDL-C < 50 mg/dL) or under lipid lowering therapy, hypertension, smoking, old (M>45, F>55 years), family history of premature CAD (M<55, F<65 years), obesity (waist: M>90, F>80 cm)] (group B).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | up to 5 years
  The composite cardiovascular (CV) outcome will be any CV events (coronary, cerebral, or peripheral vascular diseases)

SECONDARY OUTCOMES:
With at least 1 cardiovascular risk factor. | up to 5 years
  no evidence of atherosclerotic vascular diseases,with at least 1 cardiovascular risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Chau C Wu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes